CLINICAL TRIAL: NCT00788151
Title: Immunogenicity and Safety of ChimeriVax™ Tetravalent Dengue Vaccine in Healthy Children Aged 2 to 11 Years Previously Vaccinated Against Yellow Fever in Peru
Brief Title: Study of ChimeriVax™ Tetravalent Dengue Vaccine in Healthy Peruvian Children Aged 2 to 11 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD24; 2014-001711-40 (EudraCT Number)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Dengue Virus; Dengue Fever; Dengue Hemorrhagic Fever; Dengue Diseases
Keywords: Dengue virus; Dengue fever; Dengue Hemorrhagic fever; Dengue diseases; Dengue vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — ChimeriVax; Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The observer-blind design was implemented. The person who performed vaccinations knew which product was administered while neither the participant nor the Investigator in charge of safety evaluation knew which product was injected. To maintain the blind and minimize any potential bias, the control group used the same route and schedule as the study vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYD Dengue vaccine group (Experimental): Participants received three injections of the CYD Dengue vaccine at 0, 6, and 12 months. Participants were followed for 6 months after the last vaccination (up to 18 months).
  Interventions: Biological: CYD Dengue Vaccine Serotypes 1, 2, 3, and 4
- Control group (Placebo Comparator): Participants received two injections of placebo, and one injection of pneumococcal polysaccharide vaccine (Pneumo23®) at 0, 6, and 12 months, respectively. Participants were followed for 6 months after the last vaccination (up to 18 months).
  Interventions: Biological: Pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: CYD Dengue Vaccine Serotypes 1, 2, 3, and 4 — 0.5 mL, Subcutaneous (SC)
  Other Names: ChimeriVax™
  Arms: CYD Dengue vaccine group
Biological: Pneumococcal polysaccharide vaccine — 0.5 mL, SC
  Other Names: Pneumo23®
  Arms: Control group

SUMMARY:
The aim of the trial was to evaluate the use of a tetravalent vaccine, CYD dengue vaccine, against dengue disease.

Primary Objectives:

* To describe the humoral immune response to dengue before and after each vaccination with dengue vaccine in two age cohorts of children (6 to 11 years and 2 to 5 years) previously vaccinated with yellow fever (YF) vaccine.
* To evaluate the safety of each vaccination with dengue vaccine in two age cohorts of children (6 to 11 years and 2 to 5 years).
* To describe viremia after the first and second vaccinations with dengue vaccine in a subgroup of 130 randomized participants (100 participants in Dengue Vaccine Group and 30 participants in Control Group) in two age cohorts of children (6 to 11 years and 2 to 5 years).

DETAILED DESCRIPTION:
Participants were randomized to receive either three injections of CYD dengue vaccine or two injections of placebo, and one injection of a pneumococcal polysaccharide vaccine (Pneumo23®) at 0, 6, and 12 months, respectively.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 to 11 years on the day of inclusion.
* Participant in good health, based on medical history, physical examination and laboratory parameters.
* Provision of Assent Form signed by the participants (for participants >=8 years old) and Informed Consent Form signed by the parents or another legally acceptable representative (and by an independent witness for illiterate parent[s]).
* Participant and parents/legally acceptable representative able to attend all scheduled visits and to comply with all trial procedures.
* For a female participant of child-bearing potential (girls post-menarche), avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to first vaccination, until at least 4 weeks after the last vaccination.
* Documented receipt of yellow fever vaccine since at least one month before the first vaccination.

Exclusion Criteria :

* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia.
* For a female participant of child-bearing potential (girls post-menarche), known pregnancy.
* For a female participant of child-bearing potential (girls post-menarche), known pregnancy or positive pregnancy test in blood sample taken at Screening.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the trial.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of the vaccines components or history of a life-threatening reaction to the trial vaccines or to a vaccine containing any of the same substances.
* Systemic hypersensitivity to YF vaccine or history of a life-threatening reaction to YF vaccine.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Current or past alcohol abuse or drug addiction that may interfere with the participant's ability to comply with trial procedures.
* Receipt of any blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination.
* Human Immunodeficiency Virus, hepatitis B antigen, or hepatitis C seropositivity in blood sample taken at Screening.
* Clinically significant laboratory abnormalities (as determined by the Investigator) in blood sample taken at Screening.
* Known previous vaccination with pneumococcal polysaccharide vaccine.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2008-09-26 (Actual); Primary Completion 2010-02-16 (Actual); Study Completion 2010-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur SA
Locations (1):
- Chulucanas Morropon, Piura, Peru

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Crevat D. Immunogenicity and safety of tetravalent dengue vaccine in healthy Peruvian children aged 2 to 11 years, previously-vaccinated against yellow fever. "A re-emerging challenge in the Americas: opportunities for dengue research collaboration" Conference. Feb 15-18, 2011; San Juan, Puerto Rico.
- [Result] Lanata CF, Andrade T, Gil AI, Terrones C, Valladolid O, Zambrano B, Saville M, Crevat D. Immunogenicity and safety of tetravalent dengue vaccine in 2-11 year-olds previously vaccinated against yellow fever: randomized, controlled, phase II study in Piura, Peru. Vaccine. 2012 Sep 7;30(41):5935-41. doi: 10.1016/j.vaccine.2012.07.043. Epub 2012 Jul 31. PMID 22863660
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 26 September 2008 to 16 August 2010 at 1 clinical site in Peru.
Pre-assignment Details: A total of 300 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized in the study. Two participants were not vaccinated and were excluded from the Full analysis set and Safety analysis set.
Groups:
- Control Group: Participants received two injections of placebo, and 1 injection of pneumococcal polysaccharide vaccine (Pneumo23®) at 0, 6, and 12 months, respectively. Participants were followed for 6 months after the last vaccination (up to 18 months).
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Control Group
Started | 200 | 100
Received Vaccination 1 | 199 | 99
Received Vaccination 2 | 188 | 92
Received Vaccination 3 | 186 | 90
Completed | 186 | 90
Not Completed | 14 | 10
Not completed — Other adverse event | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 13 | 6
Not completed — Enrolled but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed in Full analysis set which included all the participants present at vaccination 1 and received at least 1 dose of vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Control Group | Total
Number analyzed (Participants) | 199 | 99 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.4 (2.8) | 6.4 (2.9) | 6.4 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  2 to 5 years | 100 | 50 | 150
  6 to 11 years | 99 | 49 | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 53 | 151
  Male | 101 | 46 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (Aged 2 to 11 Years) Reporting Solicited Injection-site and Systemic Reactions Following Each Injection (Inj.) With CYD Dengue Vaccine or Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Pain: Grade 3: incapacitating, unable to perform usual activities. Erythema and Swelling: Grade 3: >= 5 cm. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Fever: Grade 3: > 39.0°C; Headache, Malaise, Myalgia, and Asthenia: Grade 3: prevents daily activities.
Time Frame: Day 0 (Post-Injection) up to Day 14 after injection 1, 2 and 3
Population: Analysis was performed on Safety analysis set which included all participants who received at least 1 dose of dengue or control vaccine. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Percentage of participants
  Inj. site Pain; Post-Inj. 1 (2-11 years) | 20.6 | 17.2
  Grade 3 Inj. site Pain; Post-Inj. 1 (2-11 years) | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 1 (2-11 years) | 7.5 | 4.0
  Grade 3 Inj. site Erythema;Post-Inj.1 (2-11 years) | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 1 (2-11 years) | 5.5 | 5.1
  Grade 3 Inj. site Swelling; Post-Inj.1(2-11 years) | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Inj. site Pain; Post-Inj. 2 (2-11 years) | 19.7 | 17.4
  Grade 3 Inj. site Pain; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Inj. site Pain; Post-Inj. 2 (2-11 years) | 0.0 | 1.1
  Inj. site Erythema; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Inj. site Erythema; Post-Inj. 2 (2-11 years) | 4.3 | 1.1
  Grade 3 Inj. site Erythema;Post-Inj.2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Inj. site Erythema;Post-Inj.2 (2-11 years) | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Inj. site Swelling; Post-Inj. 2 (2-11 years) | 2.1 | 0.0
  Grade 3 Inj. site Swelling;Post-Inj.2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Inj. site Swelling;Post-Inj.2 (2-11 years) | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Inj. site Pain; Post-Inj. 3 (2-11 years) | 17.7 | 32.2
  Grade 3 Inj. site Pain; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Inj. site Pain; Post-Inj. 3 (2-11 years) | 0.5 | 2.2
  Inj. site Erythema; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Inj. site Erythema; Post-Inj. 3 (2-11 years) | 4.3 | 11.1
  Grade 3 Inj. site Erythema;Post-Inj.3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Inj. site Erythema;Post-Inj.3 (2-11 years) | 0.0 | 3.3
  Inj. site Swelling; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Inj. site Swelling; Post-Inj. 3 (2-11 years) | 3.2 | 8.9
  Grade 3 Inj. site Swelling;Post-Inj.3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Inj. site Swelling;Post-Inj.3 (2-11 years) | 0.0 | 3.3
  Fever; Post-Inj. 1 (2-11 years): number analyzed (Participants) | 198 | 99
  Fever; Post-Inj. 1 (2-11 years) | 31.3 | 10.1
  Grade 3 Fever; Post-Inj. 1 (2-11 years): number analyzed (Participants) | 198 | 99
  Grade 3 Fever; Post-Inj. 1 (2-11 years) | 3.5 | 0.0
  Headache; Post-Inj. 1 (2-11 years) | 35.7 | 16.2
  Grade 3 Headache; Post-Inj. 1 (2-11 years) | 0.5 | 0.0
  Malaise; Post-Inj. 1 (2-11 years) | 33.7 | 23.2
  Grade 3 Malaise; Post-Inj. 1 (2-11 years) | 0.5 | 0.0
  Myalgia; Post-Inj. 1 (2-11 years) | 19.1 | 13.1
  Grade 3 Myalgia; Post-Inj. 1 (2-11 years) | 0.0 | 0.0
  Asthenia; Post-Inj. 1 (2-11 years) | 13.6 | 13.1
  Grade 3 Asthenia; Post-Inj. 1 (2-11 years) | 0.5 | 0.0
  Fever; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Fever; Post-Inj. 2 (2-11 years) | 19.7 | 16.3
  Grade 3 Fever; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Fever; Post-Inj. 2 (2-11 years) | 0.5 | 0.0
  Headache; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Headache; Post-Inj. 2 (2-11 years) | 22.3 | 19.6
  Grade 3 Headache; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Headache; Post-Inj. 2 (2-11 years) | 0.5 | 1.1
  Malaise; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Malaise; Post-Inj. 2 (2-11 years) | 18.1 | 16.3
  Grade 3 Malaise; Post-Inj. 2 (All ages): number analyzed (Participants) | 188 | 92
  Grade 3 Malaise; Post-Inj. 2 (All ages) | 0.5 | 2.2
  Myalgia; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Myalgia; Post-Inj. 2 (2-11 years) | 14.9 | 10.9
  Grade 3 Myalgia; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Myalgia; Post-Inj. 2 (2-11 years) | 1.1 | 0.0
  Asthenia; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Asthenia; Post-Inj. 2 (2-11 years) | 11.2 | 7.6
  Grade 3 Asthenia; Post-Inj. 2 (2-11 years): number analyzed (Participants) | 188 | 92
  Grade 3 Asthenia; Post-Inj. 2 (2-11 years) | 0.5 | 1.1
  Fever; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 185 | 89
  Fever; Post-Inj. 3 (2-11 years) | 18.4 | 22.5
  Grade 3 Fever; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 185 | 89
  Grade 3 Fever; Post-Inj. 3 (2-11 years) | 0.0 | 3.4
  Headache; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Headache; Post-Inj. 3 (2-11 years) | 18.8 | 27.8
  Grade 3 Headache; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Headache; Post-Inj. 3 (2-11 years) | 0.0 | 3.3
  Malaise; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Malaise; Post-Inj. 3 (2-11 years) | 16.7 | 23.3
  Grade 3 Malaise; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Malaise; Post-Inj. 3 (2-11 years) | 0.0 | 2.2
  Myalgia; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Myalgia; Post-Inj. 3 (2-11 years) | 13.4 | 26.7
  Grade 3 Myalgia; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Myalgia; Post-Inj. 3 (2-11 years) | 0.0 | 2.2
  Asthenia; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Asthenia; Post-Inj. 3 (2-11 years) | 10.2 | 16.7
  Grade 3 Asthenia; Post-Inj. 3 (2-11 years): number analyzed (Participants) | 186 | 90
  Grade 3 Asthenia; Post-Inj. 3 (2-11 years) | 0.0 | 1.1

2. Primary Outcome: Percentage of Participants (Aged 2 to 5 Years) Reporting Solicited Injection-site and Systemic Reactions Following Each Injection With CYD Dengue Vaccine or Placebo
Description: as for outcome 1
Time Frame: Day 0 (Post-Injection) up to Day 14 after injection 1, 2 and 3
Population: Analysis was performed on Safety analysis set. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 100 | 50
Percentage of participants
  Inj. site Pain: Post-Inj.1 (2-5 years) | 19.0 | 16.0
  Grade 3 Inj. site Pain; Post-Inj. 1 (2-5 years) | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 1 (2-5 years) | 11.0 | 6.0
  Grade 3 Inj. site Erythema;Post-Inj. 1 (2-5 years) | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 1 (2-5 years) | 6.0 | 8.0
  Grade 3 Inj. site Swelling;Post-Inj. 1 (2-5 years) | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Inj. site Pain; Post-Inj. 2 (2-5 years) | 17.4 | 15.6
  Grade 3 Inj. site Pain; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Inj. site Pain; Post-Inj. 2 (2-5 years) | 0.0 | 2.2
  Inj. site Erythema; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Inj. site Erythema; Post-Inj. 2 (2-5 years) | 4.3 | 0.0
  Grade 3 Inj. site Erythema;Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Inj. site Erythema;Post-Inj. 2 (2-5 years) | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Inj. site Swelling; Post-Inj. 2 (2-5 years) | 2.2 | 0.0
  Grade 3 Inj. site Swelling;Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Inj. site Swelling;Post-Inj. 2 (2-5 years) | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Inj. site Pain; Post-Inj. 3 (2-5 years) | 14.4 | 23.3
  Grade 3 Inj. site Pain; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Grade 3 Inj. site Pain; Post-Inj. 3 (2-5 years) | 0.0 | 4.7
  Inj. site Erythema; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Inj. site Erythema; Post-Inj. 3 (2-5 years) | 3.3 | 9.3
  Grade 3 Inj. site Erythema;Post-Inj. 3 (2-5 years: number analyzed (Participants) | 90 | 43
  Grade 3 Inj. site Erythema;Post-Inj. 3 (2-5 years | 0.0 | 2.3
  Inj. site Swelling; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Inj. site Swelling; Post-Inj. 3 (2-5 years) | 3.3 | 7.0
  Grade 3 Inj. site Swelling;Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Grade 3 Inj. site Swelling;Post-Inj. 3 (2-5 years) | 0.0 | 2.3
  Fever; Post-Inj. 1 (2-5 years): number analyzed (Participants) | 99 | 50
  Fever; Post-Inj. 1 (2-5 years) | 36.4 | 16.0
  Grade 3 Fever; Post-Inj. 1 (2-5 years): number analyzed (Participants) | 99 | 50
  Grade 3 Fever; Post-Inj. 1 (2-5 years) | 4.0 | 0.0
  Headache; Post-Inj. 1 (2-5 years) | 23.0 | 8.0
  Grade 3 Headache; Post-Inj. 1 (2-5 years) | 1.0 | 0.0
  Malaise; Post-Inj. 1 (2-5 years) | 33.0 | 26.0
  Grade 3 Malaise; Post-Inj. 1 (2-5 years) | 1.0 | 0.0
  Myalgia; Post-Inj. 1 (2-5 years) | 12.0 | 10.0
  Grade 3 Myalgia; Post-Inj. 1 (2-5 years) | 0.0 | 0.0
  Asthenia; Post-Inj. 1 (2-5 years) | 13.0 | 12.0
  Grade 3 Asthenia; Post-Inj. 1 (2-5 years) | 1.0 | 0.0
  Fever; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Fever; Post-Inj. 2 (2-5 years) | 23.9 | 17.8
  Grade 3 Fever; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Fever; Post-Inj. 2 (2-5 years) | 0.0 | 0.0
  Headache; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Headache; Post-Inj. 2 (2-5 years) | 14.1 | 6.7
  Grade 3 Headache; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Headache; Post-Inj. 2 (2-5 years) | 0.0 | 0.0
  Malaise; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Malaise; Post-Inj. 2 (2-5 years) | 15.2 | 13.3
  Grade 3 Malaise; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Malaise; Post-Inj. 2 (2-5 years) | 1.1 | 2.2
  Myalgia; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Myalgia; Post-Inj. 2 (2-5 years) | 9.8 | 6.7
  Grade 3 Myalgia; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Myalgia; Post-Inj. 2 (2-5 years) | 1.1 | 0.0
  Asthenia; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Asthenia; Post-Inj. 2 (2-5 years) | 9.8 | 8.9
  Grade 3 Asthenia; Post-Inj. 2 (2-5 years): number analyzed (Participants) | 92 | 45
  Grade 3 Asthenia; Post-Inj. 2 (2-5 years) | 1.1 | 2.2
  Fever; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 89 | 42
  Fever; Post-Inj. 3 (2-5 years) | 16.9 | 26.2
  Grade 3 Fever; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 89 | 42
  Grade 3 Fever; Post-Inj. 3 (2-5 years) | 0.0 | 7.1
  Headache; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Headache; Post-Inj. 3 (2-5 years) | 6.7 | 18.6
  Grade 3 Headache; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Grade 3 Headache; Post-Inj. 3 (2-5 years) | 0.0 | 2.3
  Malaise; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Malaise; Post-Inj. 3 (2-5 years) | 6.7 | 23.3
  Grade 3 Malaise; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Grade 3 Malaise; Post-Inj. 3 (2-5 years) | 0.0 | 2.3
  Myalgia; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Myalgia; Post-Inj. 3 (2-5 years) | 6.7 | 20.9
  Grade 3 Myalgia; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Grade 3 Myalgia; Post-Inj. 3 (2-5 years) | 0.0 | 2.3
  Asthenia; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Asthenia; Post-Inj. 3 (2-5 years) | 4.4 | 23.3
  Grade 3 Asthenia; Post-Inj. 3 (2-5 years): number analyzed (Participants) | 90 | 43
  Grade 3 Asthenia; Post-Inj. 3 (2-5 years) | 0.0 | 2.3

3. Primary Outcome: Percentage of Participants (Aged 6 to 11 Years) Reporting Solicited Injection-site and Systemic Reactions Following Each Injection With CYD Dengue Vaccine or Placebo
Description: as for outcome 1
Time Frame: Day 0 (Post-Injection) up to Day 14 after injection 1, 2 and 3
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  Inj. site Pain; Post-Inj.1 (6-11 years) | 22.2 | 18.4
  Grade 3 Inj. site Pain; Post-Inj. 1 (6-11 years) | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 1 (6-11 years) | 4.0 | 2.0
  Grade 3 Inj. site Erythema; Post-Inj.1(6-11 years) | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 1 (6-11 years) | 5.1 | 2.0
  Grade 3 Inj. site Swelling; Post-Inj.1(6-11 years) | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Inj. site Pain; Post-Inj. 2 (6-11 years) | 21.9 | 19.1
  Grade 3 Inj. site Pain; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Inj. site Pain; Post-Inj. 2 (6-11 years) | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Inj. site Erythema; Post-Inj. 2 (6-11 years) | 4.2 | 2.1
  Grade 3 Inj. site Erythema; Post-Inj.2(6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Inj. site Erythema; Post-Inj.2(6-11 years) | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Inj. site Swelling; Post-Inj. 2 (6-11 years) | 2.1 | 0.0
  Grade 3 Inj. site Swelling; Post-Inj.2(6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Inj. site Swelling; Post-Inj.2(6-11 years) | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Inj. site Pain; Post-Inj. 3 (6-11 years) | 20.8 | 40.4
  Grade 3 Inj. site Pain; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Inj. site Pain; Post-Inj. 3 (6-11 years) | 1.0 | 0.0
  Inj. site Erythema; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Inj. site Erythema; Post-Inj. 3 (6-11 years) | 5.2 | 12.8
  Grade 3 Inj. site Erythema; Post-Inj.3(6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Inj. site Erythema; Post-Inj.3(6-11 years) | 0.0 | 4.3
  Inj. site Swelling; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Inj. site Swelling; Post-Inj. 3 (6-11 years) | 3.1 | 10.6
  Grade 3 Inj. site Swelling; Post-Inj.3(6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Inj. site Swelling; Post-Inj.3(6-11 years) | 0.0 | 4.3
  Fever; Post-Inj. 1 (6-11 years) | 26.3 | 4.1
  Grade 3 Fever; Post-Inj. 1 (6-11 years) | 3.0 | 0.0
  Headache; Post-Inj. 1 (6-11 years) | 48.5 | 24.5
  Grade 3 Headache; Post-Inj. 1 (6-11 years) | 0.0 | 0.0
  Malaise; Post-Inj. 1 (6-11 years) | 34.3 | 20.4
  Grade 3 Malaise; Post-Inj. 1 (6-11 years) | 0.0 | 0.0
  Myalgia; Post-Inj. 1 (6-11 years) | 26.3 | 16.3
  Grade 3 Myalgia; Post-Inj. 1 (6-11 years) | 0.0 | 0.0
  Asthenia; Post-Inj. 1 (6-11 years) | 14.1 | 14.3
  Grade 3 Asthenia; Post-Inj. 1 (6-11 years) | 0.0 | 0.0
  Fever; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Fever; Post-Inj. 2 (6-11 years) | 15.6 | 14.9
  Grade 3 Fever; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Fever; Post-Inj. 2 (6-11 years) | 1.0 | 0.0
  Headache; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Headache; Post-Inj. 2 (6-11 years) | 30.2 | 31.9
  Grade 3 Headache; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Headache; Post-Inj. 2 (6-11 years) | 1.0 | 2.1
  Malaise; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Malaise; Post-Inj. 2 (6-11 years) | 20.8 | 19.1
  Grade 3 Malaise; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Malaise; Post-Inj. 2 (6-11 years) | 0.0 | 2.1
  Myalgia; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Myalgia; Post-Inj. 2 (6-11 years) | 19.8 | 14.9
  Grade 3 Myalgia; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Myalgia; Post-Inj. 2 (6-11 years) | 1.0 | 0.0
  Asthenia; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Asthenia; Post-Inj. 2 (6-11 years) | 12.5 | 6.4
  Grade 3 Asthenia; Post-Inj. 2 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Asthenia; Post-Inj. 2 (6-11 years) | 0.0 | 0.0
  Fever; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Fever; Post-Inj. 3 (6-11 years) | 19.8 | 19.1
  Grade 3 Fever; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Fever; Post-Inj. 3 (6-11 years) | 0.0 | 0.0
  Headache; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Headache; Post-Inj. 3 (6-11 years) | 30.2 | 36.2
  Grade 3 Headache; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Headache; Post-Inj. 3 (6-11 years) | 0.0 | 4.3
  Malaise; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Malaise; Post-Inj. 3 (6-11 years) | 26.0 | 23.4
  Grade 3 Malaise; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Malaise; Post-Inj. 3 (6-11 years) | 0.0 | 2.1
  Myalgia; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Myalgia; Post-Inj. 3 (6-11 years) | 19.8 | 31.9
  Grade 3 Myalgia; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Myalgia; Post-Inj. 3 (6-11 years) | 0.0 | 2.1
  Asthenia; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Asthenia; Post-Inj. 3 (6-11 years) | 15.6 | 10.6
  Grade 3 Asthenia; Post-Inj. 3 (6-11 years): number analyzed (Participants) | 96 | 47
  Grade 3 Asthenia; Post-Inj. 3 (6-11 years) | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants (Aged 2 to 11 Years) Seropositive for Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity for the dengue virus serotypes was assessed by the microneutralization assay. Seropositivity was defined as a titer >=10 1/dilution.
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: Analysis was performed on Full analysis set which included all the participants present at visit 1 and who received at least one dose of vaccine. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Percentage of participants
  Dengue parental serotype 1; Pre-Inj. 1 | 29.6 | 38.4
  Dengue parental serotype 1; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  Dengue parental serotype 1; 28 days Post-Inj. 1 | 55.4 | 37.9
  Dengue parental serotype 1; Pre-Inj. 2: number analyzed (Participants) | 189 | 92
  Dengue parental serotype 1; Pre-Inj. 2 | 42.3 | 39.1
  Dengue parental serotype 1; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  Dengue parental serotype 1; 28 days Post-Inj. 2 | 98.4 | 39.1
  Dengue parental serotype 1; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  Dengue parental serotype 1; Pre-Inj. 3 | 74.7 | 41.8
  Dengue parental serotype 1; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 1; 28 days Post-Inj. 3 | 98.4 | 46.1
  Dengue parental serotype 2; Pre-Inj. 1 | 17.1 | 21.2
  Dengue parental serotype 2; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  Dengue parental serotype 2; 28 days Post-Inj. 1 | 40.4 | 21.1
  Dengue parental serotype 2; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  Dengue parental serotype 2; Pre-Inj. 2 | 32.8 | 20.4
  Dengue parental serotype 2; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  Dengue parental serotype 2; 28 days Post-Inj. 2 | 68.1 | 16.3
  Dengue parental serotype 2; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  Dengue parental serotype 2; Pre-Inj. 3 | 35.5 | 20.9
  Dengue parental serotype 2; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 2; 28 days Post-Inj. 3 | 79.0 | 20.2
  Dengue parental serotype 3; Pre-Inj. 1 | 30.7 | 38.4
  Dengue parental serotype 3; 28 days Post-Inj.1: number analyzed (Participants) | 193 | 95
  Dengue parental serotype 3; 28 days Post-Inj.1 | 68.4 | 38.9
  Dengue parental serotype 3; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  Dengue parental serotype 3; Pre-Inj. 2 | 51.9 | 39.8
  Dengue parental serotype 3; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  Dengue parental serotype 3; 28 days Post-Inj. 2 | 100.0 | 40.2
  Dengue parental serotype 3; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  Dengue parental serotype 3; Pre-Inj. 3 | 72.6 | 39.6
  Dengue parental serotype 3; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 3; 28 days Post-Inj. 3 | 98.9 | 43.8
  Dengue parental serotype 4; Pre-Inj. 1 | 14.1 | 18.2
  Dengue parental serotype 4; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  Dengue parental serotype 4; 28 days Post-Inj. 1 | 74.1 | 18.9
  Dengue parental serotype 4; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  Dengue parental serotype 4; Pre-Inj. 2 | 57.7 | 20.4
  Dengue parental serotype 4; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  Dengue parental serotype 4; 28 days Post-Inj. 2 | 97.9 | 19.6
  Dengue parental serotype 4; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  Dengue parental serotype 4; Pre-Inj. 3 | 82.8 | 18.7
  Dengue parental serotype 4; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 4; 28 days Post-Inj. 3 | 98.9 | 23.6

5. Secondary Outcome: Percentage of Participants (Aged 2 to 5 Years) Seropositive for Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: Analysis was performed on Full analysis set. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 100 | 50
Percentage of participants
  Dengue parental serotype 1; Pre-Inj. 1 | 30.0 | 32.0
  Dengue parental serotype 1; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  Dengue parental serotype 1; 28 days Post-Inj. 1 | 54.7 | 33.3
  Dengue parental serotype 1; Pre-Inj. 2: number analyzed (Participants) | 93 | 45
  Dengue parental serotype 1; Pre-Inj. 2 | 38.7 | 31.1
  Dengue parental serotype 1; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 1; 28 days Post-Inj. 2 | 97.8 | 31.1
  Dengue parental serotype 1; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  Dengue parental serotype 1; Pre-Inj. 3 | 72.2 | 36.4
  Dengue parental serotype 1; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 1; 28 days Post-Inj. 3 | 98.9 | 44.2
  Dengue parental serotype 2; Pre-Inj. 1 | 14.0 | 16.0
  Dengue parental serotype 2; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  Dengue parental serotype 2; 28 days Post-Inj. 1 | 32.6 | 16.7
  Dengue parental serotype 2; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  Dengue parental serotype 2; Pre-Inj. 2 | 29.0 | 15.2
  Dengue parental serotype 2; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 2; 28 days Post-Inj. 2 | 64.1 | 11.1
  Dengue parental serotype 2; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  Dengue parental serotype 2; Pre-Inj. 3 | 28.9 | 18.2
  Dengue parental serotype 2; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 2; 28 days Post-Inj. 3 | 77.8 | 20.9
  Dengue parental serotype 3; Pre-Inj. 1 | 28.0 | 32.0
  Dengue parental serotype 3; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  Dengue parental serotype 3; 28 days Post-Inj. 1 | 62.1 | 35.4
  Dengue parental serotype 3; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  Dengue parental serotype 3; Pre-Inj. 2 | 45.2 | 32.6
  Dengue parental serotype 3; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 3; 28 days Post-Inj. 2 | 100.0 | 33.3
  Dengue parental serotype 3; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  Dengue parental serotype 3; Pre-Inj. 3 | 70.0 | 34.1
  Dengue parental serotype 3; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 3; 28 days Post-Inj. 3 | 100.0 | 39.5
  Dengue parental serotype 4; Pre-Inj. 1 | 13.0 | 18.0
  Dengue parental serotype 4; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  Dengue parental serotype 4; 28 days Post-Inj. 1 | 74.7 | 22.9
  Dengue parental serotype 4; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  Dengue parental serotype 4; Pre-Inj. 2 | 60.2 | 17.4
  Dengue parental serotype 4; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 4; 28 days Post-Inj. 2 | 100.0 | 20.0
  Dengue parental serotype 4; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  Dengue parental serotype 4; Pre-Inj. 3 | 87.8 | 22.7
  Dengue parental serotype 4; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 4; 28 days Post-Inj. 3 | 100.0 | 27.9

6. Secondary Outcome: Percentage of Participants (Aged 6 to 11 Years) Seropositive for Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  Dengue parental serotype 1; Pre-Inj. 1 | 29.3 | 44.9
  Dengue parental serotype 1; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  Dengue parental serotype 1; 28 days Post-Inj. 1 | 56.1 | 42.6
  Dengue parental serotype 1; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 1; Pre-Inj. 2 | 45.8 | 46.8
  Dengue parental serotype 1; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 1; 28 days Post-Inj. 2 | 99.0 | 46.8
  Dengue parental serotype 1; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 1; Pre-Inj. 3 | 77.1 | 46.8
  Dengue parental serotype 1; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 1; 28 days Post-Inj. 3 | 97.9 | 47.8
  Dengue parental serotype 2; Pre-Inj. 1 | 20.2 | 26.5
  Dengue parental serotype 2; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  Dengue parental serotype 2; 28 days Post-Inj. 1 | 48.0 | 25.5
  Dengue parental serotype 2; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 2; Pre-Inj. 2 | 36.5 | 25.5
  Dengue parental serotype 2; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 2; 28 days Post-Inj. 2 | 71.9 | 21.3
  Dengue parental serotype 2; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 2; Pre-Inj. 3 | 41.7 | 23.4
  Dengue parental serotype 2; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 2; 28 days Post-Inj. 3 | 80.2 | 19.6
  Dengue parental serotype 3; Pre-Inj. 1 | 33.3 | 44.9
  Dengue parental serotype 3; 28 days Post-Inj 1: number analyzed (Participants) | 98 | 47
  Dengue parental serotype 3; 28 days Post-Inj 1 | 74.5 | 42.6
  Dengue parental serotype 3; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 3; Pre-Inj. 2 | 58.3 | 46.8
  Dengue parental serotype 3; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 3; 28 days Post-Inj. 2 | 100.0 | 46.8
  Dengue parental serotype 3; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 3; Pre-Inj. 3 | 75.0 | 44.7
  Dengue parental serotype 3; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 3; 28 days Post-Inj. 3 | 97.9 | 47.8
  Dengue parental serotype 4; Pre-Inj. 1 | 15.2 | 18.4
  Dengue parental serotype 4; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  Dengue parental serotype 4; 28 days Post-Inj. 1 | 73.5 | 14.9
  Dengue parental serotype 4; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 4; Pre-Inj. 2 | 55.2 | 23.4
  Dengue parental serotype 4; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 4; 28 days Post-Inj. 2 | 95.8 | 19.1
  Dengue parental serotype 4; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  Dengue parental serotype 4; Pre-Inj. 3 | 78.1 | 14.9
  Dengue parental serotype 4; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 4; 28 days Post-Inj. 3 | 97.9 | 19.6

7. Secondary Outcome: Percentage of Participants (Aged 2 to 11 Years) Seropositive for Dengue Virus Serotypes Before and After Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against the dengue virus serotypes was assessed by the plaque reduction neutralization test (PRNT). Seropositivity was defined as a titer >= 10 1/dilution.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: Analysis was performed on Full analysis set. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Percentage of participants
  Dengue parental serotype 1; Pre-Inj. 1: number analyzed (Participants) | 196 | 99
  Dengue parental serotype 1; Pre-Inj. 1 | 30.6 | 36.4
  Dengue parental serotype 1; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  Dengue parental serotype 1; 28 days Post-Inj. 2 | 94.7 | 39.1
  Dengue parental serotype 1; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 1; 28 days Post-Inj. 3 | 96.2 | 48.3
  Dengue parental serotype 2; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  Dengue parental serotype 2; Pre-Inj. 1 | 31.5 | 41.4
  Dengue parental serotype 2; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  Dengue parental serotype 2; 28 days Post-Inj. 2 | 97.9 | 43.5
  Dengue parental serotype 2; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 2; 28 days Post-Inj. 3 | 98.4 | 47.2
  Dengue parental serotype 3; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  Dengue parental serotype 3; Pre-Inj. 1 | 35.0 | 46.5
  Dengue parental serotype 3; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  Dengue parental serotype 3; 28 days Post-Inj. 2 | 98.9 | 51.1
  Dengue parental serotype 3; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  Dengue parental serotype 3; 28 days Post-Inj. 3 | 98.4 | 67.4
  Dengue parental serotype 4; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  Dengue parental serotype 4; Pre-Inj. 1 | 19.3 | 22.2
  Dengue parental serotype 4; 28 days Post-Inj. 2: number analyzed (Participants) | 185 | 92
  Dengue parental serotype 4; 28 days Post-Inj. 2 | 98.4 | 35.9
  Dengue parental serotype 4; 28 days Post-Inj. 3: number analyzed (Participants) | 185 | 89
  Dengue parental serotype 4; 28 days Post-Inj. 3 | 98.9 | 48.3

8. Secondary Outcome: Percentage of Participants (Aged 2 to 5 Years) Seropositive for Dengue Virus Serotypes Before and After Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity against the dengue virus serotypes was assessed by the PRNT. Seropositivity was defined as a titer >=10 1/dilution.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 100 | 50
Percentage of participants
  Dengue parental serotype 1; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  Dengue parental serotype 1; Pre-Inj. 1 | 30.3 | 30.0
  Dengue parental serotype 1; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 1; 28 days Post-Inj. 2 | 96.7 | 31.1
  Dengue parental serotype 1; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 1; 28 days Post-Inj. 3 | 97.8 | 41.9
  Dengue parental serotype 2; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  Dengue parental serotype 2; Pre-Inj. 1 | 30.3 | 38.0
  Dengue parental serotype 2; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 2; 28 days Post-Inj. 2 | 96.7 | 37.8
  Dengue parental serotype 2; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 2; 28 days Post-Inj. 3 | 100.0 | 44.2
  Dengue parental serotype 3; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  Dengue parental serotype 3; Pre-Inj. 1 | 35.4 | 38.0
  Dengue parental serotype 3; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  Dengue parental serotype 3; 28 days Post-Inj. 2 | 98.9 | 53.3
  Dengue parental serotype 3; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 3; 28 days Post-Inj. 3 | 98.9 | 65.1
  Dengue parental serotype 4; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  Dengue parental serotype 4; Pre-Inj. 1 | 16.2 | 22.0
  Dengue parental serotype 4; 28 days Post-Inj. 2: number analyzed (Participants) | 90 | 45
  Dengue parental serotype 4; 28 days Post-Inj. 2 | 97.8 | 35.6
  Dengue parental serotype 4; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  Dengue parental serotype 4; 28 days Post-Inj. 3 | 100.0 | 46.5

9. Secondary Outcome: Percentage of Participants (Aged 6 to 11 Years) Seropositive for Dengue Virus Serotypes Before and After Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 8
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  Dengue parental serotype 1; Pre-Inj. 1: number analyzed (Participants) | 97 | 49
  Dengue parental serotype 1; Pre-Inj. 1 | 30.9 | 42.9
  Dengue parental serotype 1; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  Dengue parental serotype 1; 28 days Post-Inj. 2 | 92.6 | 46.8
  Dengue parental serotype 1; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 1; 28 days Post-Inj. 3 | 94.8 | 54.3
  Dengue parental serotype 2; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  Dengue parental serotype 2; Pre-Inj. 1 | 32.7 | 44.9
  Dengue parental serotype 2; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  Dengue parental serotype 2; 28 days Post-Inj. 2 | 98.9 | 48.9
  Dengue parental serotype 2; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 2; 28 days Post-Inj. 3 | 96.9 | 50.0
  Dengue parental serotype 3; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  Dengue parental serotype 3; Pre-Inj. 1 | 34.7 | 55.1
  Dengue parental serotype 3; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  Dengue parental serotype 3; 28 days Post-Inj. 2 | 98.9 | 48.9
  Dengue parental serotype 3; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  Dengue parental serotype 3; 28 days Post-Inj. 3 | 97.9 | 69.6
  Dengue parental serotype 4; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  Dengue parental serotype 4; Pre-Inj. 1 | 22.4 | 22.4
  Dengue parental serotype 4; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  Dengue parental serotype 4; 28 days Post-Inj. 2 | 98.9 | 36.2
  Dengue parental serotype 4; 28 days Post-Inj. 3: number analyzed (Participants) | 95 | 46
  Dengue parental serotype 4; 28 days Post-Inj. 3 | 97.9 | 50.0

10. Secondary Outcome: Percentage of Participants (Aged 2 to 11 Years) Seropositive for at Least One, Two, Three or Four Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Percentage of participants
  At least 1 positive serotype; Pre-Inj. 1 | 32.2 | 40.4
  At least 1 positive serotype; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  At least 1 positive serotype; 28 days Post-Inj. 1 | 80.8 | 40.0
  At least 1 positive serotype; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  At least 1 positive serotype; Pre-Inj. 2 | 69.8 | 40.9
  At least 1 positive serotype; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  At least 1 positive serotype; 28 days Post-Inj. 2 | 100.0 | 42.4
  At least 1 positive serotype; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  At least 1 positive serotype; Pre-Inj. 3 | 88.7 | 42.9
  At least 1 positive serotype; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  At least 1 positive serotype; 28 days Post-Inj. 3 | 98.9 | 48.3
  At least 2 positive serotypes; Pre-Inj. 1 | 29.1 | 38.4
  At least 2 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  At least 2 positive serotypes; 28 days Post-Inj. 1 | 66.8 | 38.9
  At least 2 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  At least 2 positive serotypes; Pre-Inj. 2 | 49.2 | 39.8
  At least 2 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  At least 2 positive serotypes; 28 days Post-Inj. 2 | 100.0 | 40.2
  At least 2 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  At least 2 positive serotypes; Pre-Inj. 3 | 75.3 | 39.6
  At least 2 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  At least 2 positive serotypes; 28 days Post-Inj. 3 | 98.9 | 43.8
  At least 3 positive serotypes; Pre-Inj. 1 | 19.6 | 24.2
  At least 3 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  At least 3 positive serotypes; 28 days Post-Inj. 1 | 52.8 | 25.3
  At least 3 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  At least 3 positive serotypes; Pre-Inj. 2 | 38.1 | 22.6
  At least 3 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  At least 3 positive serotypes; 28 days Post-Inj. 2 | 98.4 | 21.7
  At least 3 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  At least 3 positive serotypes; Pre-Inj. 3 | 67.7 | 25.3
  At least 3 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  At least 3 positive serotypes; 28 days Post-Inj. 3 | 98.4 | 25.8
  All 4 positive serotypes; Pre-Inj. 1 | 10.6 | 13.1
  All 4 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 193 | 95
  All 4 positive serotypes; 28 days Post-Inj. 1 | 37.8 | 12.6
  All 4 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 189 | 93
  All 4 positive serotypes; Pre-Inj. 2 | 27.5 | 16.1
  All 4 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 188 | 92
  All 4 positive serotypes; 28 days Post-Inj. 2 | 66.0 | 10.9
  All 4 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 186 | 91
  All 4 positive serotypes; Pre-Inj. 3 | 33.9 | 13.2
  All 4 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  All 4 positive serotypes; 28 days Post-Inj. 3 | 79.0 | 15.7

11. Secondary Outcome: Percentage of Participants (Aged 2 to 5 Years) Seropositive for at Least One, Two, Three or Four Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine or Placebo
Description: Seropositivity for the dengue virus serotypes was assessed by the microneutralization assay. Seropositivity was defined as a titer >= 10 1/dilution.
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 100 | 50
Percentage of participants
  At least 1 positive serotype; Pre-Inj. 1 | 31.0 | 34.0
  At least 1 positive serotype; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  At least 1 positive serotype; 28 days Post-Inj. 1 | 78.9 | 35.4
  At least 1 positive serotype; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  At least 1 positive serotype; Pre-Inj. 2 | 67.7 | 32.6
  At least 1 positive serotype; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  At least 1 positive serotype; 28 days Post-Inj. 2 | 100.0 | 33.3
  At least 1 positive serotype; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  At least 1 positive serotype; Pre-Inj. 3 | 90.0 | 36.4
  At least 1 positive serotype; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  At least 1 positive serotype; 28 days Post-Inj. 3 | 100.0 | 44.2
  At least 2 positive serotypes; Pre-Inj. 1 | 28.0 | 32.0
  At least 2 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  At least 2 positive serotypes; 28 days Post-Inj. 1 | 65.3 | 35.4
  At least 2 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  At least 2 positive serotypes; Pre-Inj. 2 | 46.2 | 32.6
  At least 2 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  At least 2 positive serotypes; 28 days Post-Inj. 2 | 100.0 | 33.3
  At least 2 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  At least 2 positive serotypes; Pre-Inj. 3 | 75.6 | 34.1
  At least 2 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  At least 2 positive serotypes; 28 days Post-Inj. 3 | 100.0 | 39.5
  At least 3 positive serotypes; Pre-Inj. 1 | 17.0 | 24.0
  At least 3 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  At least 3 positive serotypes; 28 days Post-Inj. 1 | 48.4 | 27.1
  At least 3 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  At least 3 positive serotypes; Pre-Inj. 2 | 33.3 | 19.6
  At least 3 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  At least 3 positive serotypes; 28 days Post-Inj. 2 | 98.9 | 20.0
  At least 3 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  At least 3 positive serotypes; Pre-Inj. 3 | 65.6 | 27.3
  At least 3 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  At least 3 positive serotypes; 28 days Post-Inj. 3 | 98.9 | 30.2
  All 4 positive serotypes; Pre-Inj. 1 | 9.0 | 8.0
  All 4 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 95 | 48
  All 4 positive serotypes; 28 days Post-Inj. 1 | 31.6 | 10.4
  All 4 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 93 | 46
  All 4 positive serotypes; Pre-Inj. 2 | 25.8 | 10.9
  All 4 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  All 4 positive serotypes; 28 days Post-Inj. 2 | 63.0 | 8.9
  All 4 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 90 | 44
  All 4 positive serotypes; Pre-Inj. 3 | 27.8 | 13.6
  All 4 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  All 4 positive serotypes; 28 days Post-Inj. 3 | 77.8 | 18.6

12. Secondary Outcome: Percentage of Participants (Aged 6 to 11 Years) Seropositive for at Least One, Two, Three or Four Dengue Virus Serotypes Before and After Each Vaccination With CYD Dengue Vaccine
Description: as for outcome 4
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  At least 1 positive serotype; Pre-Inj. 1 | 33.3 | 46.9
  At least 1 positive serotype; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  At least 1 positive serotype; 28 days Post-Inj. 1 | 82.7 | 44.7
  At least 1 positive serotype; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  At least 1 positive serotype; Pre-Inj. 2 | 71.9 | 48.9
  At least 1 positive serotype; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  At least 1 positive serotype; 28 days Post-Inj. 2 | 100.0 | 51.1
  At least 1 positive serotype; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  At least 1 positive serotype; Pre-Inj. 3 | 87.5 | 48.9
  At least 1 positive serotype; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  At least 1 positive serotype; 28 days Post-Inj. 3 | 97.9 | 52.2
  At least 2 positive serotypes; Pre-Inj. 1 | 30.3 | 44.9
  At least 2 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  At least 2 positive serotypes; 28 days Post-Inj. 1 | 68.4 | 42.6
  At least 2 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  At least 2 positive serotypes; Pre-Inj. 2 | 52.1 | 46.8
  At least 2 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  At least 2 positive serotypes; 28 days Post-Inj. 2 | 100.0 | 46.8
  At least 2 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  At least 2 positive serotypes; Pre-Inj. 3 | 75.0 | 44.7
  At least 2 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  At least 2 positive serotypes; 28 days Post-Inj. 3 | 97.9 | 47.8
  At least 3 positive serotypes; Pre-Inj. 1 | 22.2 | 24.5
  At least 3 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  At least 3 positive serotypes; 28 days Post-Inj. 1 | 57.1 | 23.4
  At least 3 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  At least 3 positive serotypes; Pre-Inj. 2 | 42.7 | 25.5
  At least 3 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  At least 3 positive serotypes; 28 days Post-Inj. 2 | 97.9 | 23.4
  At least 3 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  At least 3 positive serotypes; Pre-Inj. 3 | 69.8 | 23.4
  At least 3 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  At least 3 positive serotypes; 28 days Post-Inj. 3 | 97.9 | 21.7
  All 4 positive serotypes; Pre-Inj. 1 | 12.1 | 18.4
  All 4 positive serotypes; 28 days Post-Inj. 1: number analyzed (Participants) | 98 | 47
  All 4 positive serotypes; 28 days Post-Inj. 1 | 43.9 | 14.9
  All 4 positive serotypes; Pre-Inj. 2: number analyzed (Participants) | 96 | 47
  All 4 positive serotypes; Pre-Inj. 2 | 29.2 | 21.3
  All 4 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 96 | 47
  All 4 positive serotypes; 28 days Post-Inj. 2 | 68.8 | 12.8
  All 4 positive serotypes; Pre-Inj. 3: number analyzed (Participants) | 96 | 47
  All 4 positive serotypes; Pre-Inj. 3 | 39.6 | 12.8
  All 4 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  All 4 positive serotypes; 28 days Post-Inj. 3 | 80.2 | 13.0

13. Secondary Outcome: Percentage of Participants (Aged 2 to 11 Years) Seropositive for at Least One, Two, Three or Four Dengue Virus Serotypes Before and After Vaccination With CYD Dengue Vaccine
Description: as for outcome 8
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Percentage of participants
  At least 1 positive serotype; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  At least 1 positive serotype; Pre-Inj. 1 | 37.6 | 48.5
  At least 1 positive serotype; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  At least 1 positive serotype; 28 days Post-Inj. 2 | 100.0 | 57.6
  At least 1 positive serotype; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  At least 1 positive serotype; 28 days Post-Inj. 3 | 99.5 | 73.0
  At least 2 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  At least 2 positive serotypes; Pre-Inj. 1 | 31.5 | 41.4
  At least 2 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  At least 2 positive serotypes; 28 days Post-Inj. 2 | 99.5 | 41.3
  At least 2 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  At least 2 positive serotypes; 28 days Post-Inj. 3 | 99.5 | 52.8
  At least 3 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  At least 3 positive serotypes; Pre-Inj. 1 | 29.9 | 37.4
  At least 3 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  At least 3 positive serotypes; 28 days Post-Inj. 2 | 98.4 | 41.3
  At least 3 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  At least 3 positive serotypes; 28 days Post-Inj. 3 | 98.4 | 46.1
  All 4 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 197 | 99
  All 4 positive serotypes; Pre-Inj. 1 | 17.3 | 19.2
  All 4 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 187 | 92
  All 4 positive serotypes; 28 days Post-Inj. 2 | 90.9 | 29.3
  All 4 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 186 | 89
  All 4 positive serotypes; 28 days Post-Inj. 3 | 94.1 | 39.3

14. Secondary Outcome: Percentage of Participants (Aged 2 to 5 Years) Seropositive for at Least One, Two, Three or Four Dengue Virus Serotypes Before and After Vaccination With CYD Dengue Vaccine
Description: Seropositivity against the dengue virus serotypes was assessed by the PRNT. Seropositivity was defined as a titer >= 10 1/dilution.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 100 | 50
Percentage of participants
  At least 1 positive serotype; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  At least 1 positive serotype; Pre-Inj. 1 | 39.4 | 42.0
  At least 1 positive serotype; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  At least 1 positive serotype; 28 days Post-Inj. 2 | 100.0 | 64.4
  At least 1 positive serotype; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  At least 1 positive serotype; 28 days Post-Inj. 3 | 100.0 | 74.4
  At least 2 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  At least 2 positive serotypes; Pre-Inj. 1 | 30.3 | 36.0
  At least 2 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  At least 2 positive serotypes; 28 days Post-Inj. 2 | 100.0 | 33.3
  At least 2 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  At least 2 positive serotypes; 28 days Post-Inj. 3 | 100.0 | 44.2
  At least 3 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  At least 3 positive serotypes; Pre-Inj. 1 | 28.3 | 34.0
  At least 3 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  At least 3 positive serotypes; 28 days Post-Inj. 2 | 97.8 | 33.3
  At least 3 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  At least 3 positive serotypes; 28 days Post-Inj. 3 | 100 | 41.9
  All 4 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 99 | 50
  All 4 positive serotypes; Pre-Inj. 1 | 14.1 | 16.0
  All 4 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 92 | 45
  All 4 positive serotypes; 28 days Post-Inj. 2 | 90.2 | 26.7
  All 4 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 90 | 43
  All 4 positive serotypes; 28 days Post-Inj. 3 | 96.7 | 37.2

15. Secondary Outcome: Percentage of Participants (Aged 6 to 11 Years) Seropositive for at Least One, Two, Three or Four Dengue Virus Serotypes Before and After Vaccination With CYD Dengue Vaccine
Description: as for outcome 8
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  At least 1 positive serotype; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  At least 1 positive serotype; Pre-Inj. 1 | 35.7 | 55.1
  At least 1 positive serotype; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  At least 1 positive serotype; 28 days Post-Inj. 2 | 100.0 | 51.1
  At least 1 positive serotype; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  At least 1 positive serotype; 28 days Post-Inj. 3 | 99.0 | 71.7
  At least 2 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  At least 2 positive serotypes; Pre-Inj. 1 | 32.7 | 46.9
  At least 2 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  At least 2 positive serotypes; 28 days Post-Inj. 2 | 98.9 | 48.9
  At least 2 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  At least 2 positive serotypes; 28 days Post-Inj. 3 | 99.0 | 60.9
  At least 3 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  At least 3 positive serotypes; Pre-Inj. 1 | 31.6 | 40.8
  At least 3 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  At least 3 positive serotypes; 28 days Post-Inj. 2 | 98.9 | 48.9
  At least 3 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  At least 3 positive serotypes; 28 days Post-Inj. 3 | 96.9 | 50.0
  All 4 positive serotypes; Pre-Inj. 1: number analyzed (Participants) | 98 | 49
  All 4 positive serotypes; Pre-Inj. 1 | 20.4 | 22.4
  All 4 positive serotypes; 28 days Post-Inj. 2: number analyzed (Participants) | 95 | 47
  All 4 positive serotypes; 28 days Post-Inj. 2 | 91.6 | 31.9
  All 4 positive serotypes; 28 days Post-Inj. 3: number analyzed (Participants) | 96 | 46
  All 4 positive serotypes; 28 days Post-Inj. 3 | 91.7 | 41.3

16. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Dengue Virus Serotype in Dengue-Immune Participants Before and After Injection With CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against parental dengue virus serotypes were assessed by the PRNT. GMTs values are reported for all participants in each reporting arm and also separately for participants with age 2-5 years and 6-11 years.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 2 and 3
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Titers (1/dilution)
  Serotype 1; Pre-Inj. 1, All: number analyzed (Participants) | 196 | 99
  Serotype 1; Pre-Inj. 1, All | 17.4 [13.0 to 23.2] | 22.8 [14.9 to 34.8]
  Serotype 1; 28 days Post-Inj. 2, All: number analyzed (Participants) | 187 | 92
  Serotype 1; 28 days Post-Inj. 2, All | 125 [98.5 to 159] | 26.4 [16.7 to 41.8]
  Serotype 1; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 1; 28 days Post-Inj. 3, All | 179 [143 to 224] | 38.1 [23.4 to 62.1]
  Serotype 2; Pre-Inj. 1, All: number analyzed (Participants) | 197 | 99
  Serotype 2; Pre-Inj. 1, All | 14.4 [11.2 to 18.3] | 18.2 [12.8 to 25.8]
  Serotype 2; 28 days Post-Inj. 2, All: number analyzed (Participants) | 187 | 92
  Serotype 2; 28 days Post-Inj. 2, All | 151 [128 to 178] | 17.3 [12.5 to 23.9]
  Serotype 2; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 2; 28 days Post-Inj. 3, All | 178 [152 to 207] | 21.6 [14.8 to 31.5]
  Serotype 3; Pre-Inj. 1, All: number analyzed (Participants) | 197 | 99
  Serotype 3; Pre-Inj. 1, All | 16.4 [12.7 to 21.2] | 21.8 [15.2 to 31.3]
  Serotype 3; 28 days Post-Inj. 2, All: number analyzed (Participants) | 187 | 92
  Serotype 3; 28 days Post-Inj. 2, All | 155 [129 to 186] | 26.6 [18.1 to 39.0]
  Serotype 3; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 3; 28 days Post-Inj. 3, All | 190 [162 to 224] | 36.2 [25.1 to 52.0]
  Serotype 4; Pre-Inj. 1, All: number analyzed (Participants) | 197 | 99
  Serotype 4; Pre-Inj. 1, All | 8.12 [6.91 to 9.54] | 8.94 [6.97 to 11.5]
  Serotype 4; 28 days Post-Inj. 2, All: number analyzed (Participants) | 185 | 92
  Serotype 4; 28 days Post-Inj. 2, All | 144 [126 to 166] | 12.8 [9.50 to 17.2]
  Serotype 4; 28 days Post-Inj. 3, All: number analyzed (Participants) | 185 | 89
  Serotype 4; 28 days Post-Inj. 3, All | 184 [159 to 212] | 16.7 [12.2 to 22.8]
  Serotype 1; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 99 | 50
  Serotype 1; Pre-Inj. 1, 2-5 years | 16.4 [11.1 to 24.3] | 16.2 [9.47 to 27.5]
  Serotype 1; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 1; 28 days Post-Inj. 2, 2-5 years | 135 [97.2 to 187] | 19.0 [10.1 to 35.7]
  Serotype 1; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 1; 28 days Post-Inj. 3, 2-5 years | 205 [149 to 282] | 31.3 [14.9 to 65.9]
  Serotype 2; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 99 | 50
  Serotype 2; Pre-Inj. 1, 2-5 years | 11.8 [8.94 to 15.6] | 13.9 [9.31 to 20.6]
  Serotype 2; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 2; 28 days Post-Inj. 2, 2-5 years | 135 [109 to 168] | 13.2 [8.80 to 19.9]
  Serotype 2; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 2; 28 days Post-Inj. 3, 2-5 years | 195 [163 to 234] | 21.8 [12.1 to 39.2]
  Serotype 3; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 99 | 50
  Serotype 3; Pre-Inj. 1, 2-5 years | 16.2 [11.2 to 23.4] | 16.7 [10.2 to 27.4]
  Serotype 3; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 3; 28 days Post-Inj. 2, 2-5 years | 171 [131 to 224] | 26.5 [15.4 to 45.7]
  Serotype 3; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 3; 28 days Post-Inj. 3, 2-5 years | 214 [169 to 270] | 35.0 [20.3 to 60.6]
  Serotype 4; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 99 | 50
  Serotype 4; Pre-Inj. 1, 2-5 years | 7.76 [6.20 to 9.70] | 9.02 [6.27 to 13.0]
  Serotype 4; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 90 | 45
  Serotype 4; 28 days Post-Inj. 2, 2-5 years | 165 [134 to 203] | 14.4 [8.83 to 23.6]
  Serotype 4; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 4; 28 days Post-Inj. 3, 2-5 years | 223 [181 to 276] | 18.7 [11.2 to 31.4]
  Serotype 1; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 97 | 49
  Serotype 1; Pre-Inj. 1, 6-11 years | 18.4 [12.0 to 28.4] | 32.3 [16.6 to 63.1]
  Serotype 1; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 95 | 47
  Serotype 1; 28 days Post-Inj. 2, 6-11 years | 116 [81.7 to 165] | 36.2 [18.5 to 71.0]
  Serotype 1; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 1; 28 days Post-Inj. 3, 6-11 years | 157 [115 to 216] | 45.8 [23.6 to 88.8]
  Serotype 2; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 49
  Serotype 2; Pre-Inj. 1, 6-11 years | 17.5 [11.6 to 26.3] | 24.0 [13.4 to 43.1]
  Serotype 2; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 95 | 47
  Serotype 2; 28 days Post-Inj. 2, 6-11 years | 168 [130 to 216] | 22.3 [13.4 to 37.0]
  Serotype 2; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 2; 28 days Post-Inj. 3, 6-11 years | 163 [127 to 208] | 21.4 [12.9 to 35.6]
  Serotype 3; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 49
  Serotype 3; Pre-Inj. 1, 6-11 years | 16.6 [11.5 to 24.0] | 28.6 [16.7 to 48.7]
  Serotype 3; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 95 | 47
  Serotype 3; 28 days Post-Inj. 2, 6-11 years | 141 [109 to 182] | 26.6 [15.1 to 46.8]
  Serotype 3; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 3; 28 days Post-Inj. 3, 6-11 years | 171 [137 to 213] | 37.3 [22.5 to 61.6]
  Serotype 4; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 49
  Serotype 4; Pre-Inj. 1, 6-11 years | 8.50 [6.72 to 10.8] | 8.87 [6.21 to 12.6]
  Serotype 4; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 95 | 47
  Serotype 4; 28 days Post-Inj. 2, 6-11 years | 127 [106 to 153] | 11.4 [7.96 to 16.3]
  Serotype 4; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 95 | 46
  Serotype 4; 28 days Post-Inj. 3, 6-11 years | 152 [126 to 184] | 15.0 [10.2 to 22.0]

17. Secondary Outcome: Percentage of Participants Seropositive for Yellow Fever Antibodies Before and Following First Injection With CYD Dengue Vaccine or Placebo
Description: Seropositivity for yellow fever was assessed by the PRNT. Seropositivity was defined as a titer >=10 1/dilution. Percentage values are reported for all participants in each reporting arm and also separately for participants with age 2-5 years and 6-11 years.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 1
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Percentage of participants
  Pre-Inj. 1; All participants | 81.4 | 83.8
  28 days Post-Inj. 1; All participants: number analyzed (Participants) | 192 | 95
  28 days Post-Inj. 1; All participants | 86.5 | 83.2
  Pre-Inj. 1; 2-5 years: number analyzed (Participants) | 100 | 50
  Pre-Inj. 1; 2-5 years | 68.0 | 74.0
  28 days Post-Inj. 1; 2-5 years: number analyzed (Participants) | 94 | 48
  28 days Post-Inj. 1; 2-5 years | 76.6 | 72.9
  Pre-Inj. 1; 6-11 years: number analyzed (Participants) | 99 | 49
  Pre-Inj. 1; 6-11 years | 94.9 | 93.9
  28 days Post-Inj. 1; 6-11 years: number analyzed (Participants) | 98 | 47
  28 days Post-Inj. 1; 6-11 years | 95.9 | 93.6

18. Secondary Outcome: GMTs of Antibodies Against Yellow Fever Virus Before and Following First Injection With CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against yellow fever virus were assessed by the PRNT. GMTs values are reported for all participants in each reporting arm and also separately for participants with age 2-5 years and 6-11 years.
Time Frame: Pre-Injection 1 and 28 days Post-Injection 1
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Titers (1/dilution)
  Pre-Inj. 1; All participants | 32.3 [26.5 to 39.4] | 36.0 [27.1 to 47.7]
  28 days Post-Inj. 1; All participants: number analyzed (Participants) | 192 | 95
  28 days Post-Inj. 1; All participants | 43.7 [36.1 to 52.8] | 36.0 [27.3 to 47.3]
  Pre-Inj. 1; 2-5 years: number analyzed (Participants) | 100 | 50
  Pre-Inj. 1; 2-5 years | 15.9 [12.3 to 20.6] | 20.5 [13.7 to 30.7]
  28 days Post-Inj. 1; 2-5 years: number analyzed (Participants) | 94 | 48
  28 days Post-Inj. 1; 2-5 years | 22.4 [17.5 to 28.7] | 21.2 [14.4 to 31.1]
  Pre-Inj. 1; 6-11 years: number analyzed (Participants) | 99 | 49
  Pre-Inj. 1; 6-11 years | 66.1 [52.8 to 82.9] | 63.9 [45.8 to 89.2]
  28 days Post-Inj. 1; 6-11 years: number analyzed (Participants) | 98 | 47
  28 days Post-Inj. 1; 6-11 years | 82.9 [66.2 to 104] | 61.8 [44.0 to 86.7]

19. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Before and Following Injection With CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against parental dengue virus serotypes were assessed by the microneutralization assay. GMTs values are reported for all participants in each reporting arm and also separately for participants with age 2-5 years and 6-11 years.
Time Frame: Pre-Injection 1, 2, 3 and 28 days Post-Injection 1, 2 and 3
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 199 | 99
Titers (1/dilution)
  Serotype 1; Pre-Inj. 1, All | 18.8 [13.8 to 25.6] | 23.9 [15.5 to 36.9]
  Serotype 1; 28 days Post-Inj.1, All: number analyzed (Participants) | 193 | 95
  Serotype 1; 28 days Post-Inj.1, All | 43.1 [30.0 to 61.9] | 22.8 [14.8 to 35.1]
  Serotype 1; Pre-Inj. 2, All: number analyzed (Participants) | 189 | 92
  Serotype 1; Pre-Inj. 2, All | 29.2 [20.5 to 41.7] | 26.0 [16.2 to 41.5]
  Serotype 1; 28 days Post-Inj. 2, All: number analyzed (Participants) | 188 | 92
  Serotype 1; 28 days Post-Inj. 2, All | 214 [171 to 266] | 26.1 [16.3 to 42.0]
  Serotype 1; Pre-Inj. 3, All: number analyzed (Participants) | 186 | 91
  Serotype 1; Pre-Inj. 3, All | 64.1 [46.1 to 89.2] | 28.9 [17.7 to 49.3]
  Serotype 1; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 1; 28 days Post-Inj. 3, All | 254 [203 to 318] | 35.3 [21.2 to 58.7]
  Serotype 2; Pre-Inj. 1, All | 7.55 [6.50 to 8.78] | 7.76 [6.31 to 9.53]
  Serotype 2; 28 days Post-Inj.1, All: number analyzed (Participants) | 193 | 95
  Serotype 2; 28 days Post-Inj.1, All | 15.5 [12.4 to 19.4] | 7.51 [6.19 to 9.12]
  Serotype 2; Pre-Inj. 2, All: number analyzed (Participants) | 189 | 93
  Serotype 2; Pre-Inj. 2, All | 11.6 [9.52 to 14.1] | 7.32 [6.06 to 8.84]
  Serotype 2; 28 days Post-Inj. 2, All: number analyzed (Participants) | 188 | 92
  Serotype 2; 28 days Post-Inj. 2, All | 21.4 [17.6 to 25.9] | 6.99 [5.82 to 8.39]
  Serotype 2; Pre-Inj. 3, All: number analyzed (Participants) | 186 | 91
  Serotype 2; Pre-Inj. 3, All | 11.4 [9.39 to 13.8] | 7.26 [6.01 to 8.78]
  Serotype 2; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 2; 28 days Post-Inj. 3, All | 22.3 [18.9 to 26.4] | 7.73 [6.24 to 9.58]
  Serotype 3; Pre-Inj. 1, All | 13.1 [10.3 to 16.5] | 16.3 [11.6 to 22.8]
  Serotype 3; 28 days Post-Inj.1, All: number analyzed (Participants) | 193 | 95
  Serotype 3; 28 days Post-Inj.1, All | 41.4 [30.9 to 55.4] | 15.3 [11.0 to 21.3]
  Serotype 3; Pre-Inj. 2, All: number analyzed (Participants) | 189 | 93
  Serotype 3; Pre-Inj. 2, All | 22.6 [17.3 to 29.5] | 15.4 [11.2 to 21.2]
  Serotype 3; 28 days Post-Inj. 2, All: number analyzed (Participants) | 188 | 92
  Serotype 3; 28 days Post-Inj. 2, All | 128 [108 to 150] | 15.5 [11.2 to 21.5]
  Serotype 3; Pre-Inj. 3, All: number analyzed (Participants) | 186 | 91
  Serotype 3; Pre-Inj. 3, All | 31.0 [24.3 to 39.6] | 14.0 [10.3 to 19.0]
  Serotype 3; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 3; 28 days Post-Inj. 3, All | 99.2 [84.8 to 116] | 16.0 [11.5 to 22.2]
  Serotype 4; Pre-Inj. 1, All | 7.52 [6.37 to 8.87] | 8.08 [6.39 to 10.2]
  Serotype 4; 28 days Post-Inj.1, All: number analyzed (Participants) | 193 | 95
  Serotype 4; 28 days Post-Inj.1, All | 87.9 [65.4 to 118] | 7.84 [6.25 to 9.83]
  Serotype 4; Pre-Inj. 2, All: number analyzed (Participants) | 189 | 93
  Serotype 4; Pre-Inj. 2, All | 21.3 [16.9 to 26.8] | 7.73 [6.27 to 9.53]
  Serotype 4; 28 days Post-Inj. 2, All: number analyzed (Participants) | 188 | 92
  Serotype 4; 28 days Post-Inj. 2, All | 158 [134 to 186] | 7.81 [6.27 to 9.74]
  Serotype 4; Pre-Inj. 3, All: number analyzed (Participants) | 186 | 91
  Serotype 4; Pre-Inj. 3, All | 39.2 [31.7 to 48.5] | 7.49 [6.06 to 9.26]
  Serotype 4; 28 days Post-Inj. 3, All: number analyzed (Participants) | 186 | 89
  Serotype 4; 28 days Post-Inj. 3, All | 147 [126 to 172] | 8.54 [6.71 to 10.9]
  Serotype 1; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 100 | 50
  Serotype 1; Pre-Inj. 1, 2-5 years | 20.3 [12.9 to 32.0] | 18.6 [10.4 to 33.4]
  Serotype 1; 28 days Post-Inj. 1, 2-5 years: number analyzed (Participants) | 95 | 48
  Serotype 1; 28 days Post-Inj. 1, 2-5 years | 44.8 [25.9 to 77.3] | 19.6 [10.6 to 36.1]
  Serotype 1; Pre-Inj. 2, 2-5 years: number analyzed (Participants) | 93 | 45
  Serotype 1; Pre-Inj. 2, 2-5 years | 31.3 [18.1 to 53.9] | 19.7 [10.1 to 38.2]
  Serotype 1; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 1; 28 days Post-Inj. 2, 2-5 years | 281 [204 to 386] | 20.9 [10.5 to 41.7]
  Serotype 1; Pre-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 44
  Serotype 1; Pre-Inj. 3, 2-5 years | 65.2 [39.6 to 107] | 22.1 [11.0 to 44.5]
  Serotype 1; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 1; 28 days Post-Inj. 3, 2-5 years | 315 [228 to 436] | 35.9 [16.4 to 78.6]
  Serotype 2; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 100 | 50
  Serotype 2; Pre-Inj. 1, 2-5 years | 6.66 [5.63 to 7.88] | 6.48 [5.30 to 7.92]
  Serotype 2; 28 days Post-Inj. 1, 2-5 years: number analyzed (Participants) | 95 | 48
  Serotype 2; 28 days Post-Inj. 1, 2-5 years | 12.7 [9.35 to 17.3] | 6.73 [5.39 to 8.41]
  Serotype 2; Pre-Inj. 2, 2-5 years: number analyzed (Participants) | 93 | 46
  Serotype 2; Pre-Inj. 2, 2-5 years | 10.1 [7.85 to 12.9] | 6.28 [5.19 to 7.61]
  Serotype 2; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 2; 28 days Post-Inj. 2, 2-5 years | 17.1 [13.4 to 21.8] | 6.13 [5.06 to 7.44]
  Serotype 2; Pre-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 44
  Serotype 2; Pre-Inj. 3, 2-5 years | 9.03 [7.17 to 11.4] | 6.68 [5.37 to 8.32]
  Serotype 2; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 2; 28 days Post-Inj. 3, 2-5 years | 19.7 [15.9 to 24.5] | 7.93 [5.76 to 10.9]
  Serotype 3; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 100 | 50
  Serotype 3; Pre-Inj. 1, 2-5 years | 11.8 [8.54 to 16.4] | 12.2 [8.00 to 18.7]
  Serotype 3; 28 days Post-Inj. 1, 2-5 years: number analyzed (Participants) | 95 | 48
  Serotype 3; 28 days Post-Inj. 1, 2-5 years | 37.4 [23.9 to 58.3] | 12.9 [8.39 to 20.0]
  Serotype 3; Pre-Inj. 2, 2-5 years: number analyzed (Participants) | 93 | 46
  Serotype 3; Pre-Inj. 2, 2-5 years | 19.8 [13.4 to 29.4] | 12.3 [7.92 to 19.0]
  Serotype 3; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 3; 28 days Post-Inj. 2, 2-5 years | 129 [104 to 160] | 12.6 [8.01 to 19.7]
  Serotype 3; Pre-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 44
  Serotype 3; Pre-Inj. 3, 2-5 years | 26.7 [18.7 to 38.2] | 12.2 [7.85 to 19.1]
  Serotype 3; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 3; 28 days Post-Inj. 3, 2-5 years | 108 [86.9 to 135] | 15.3 [9.29 to 25.2]
  Serotype 4; Pre-Inj. 1, 2-5 years: number analyzed (Participants) | 100 | 50
  Serotype 4; Pre-Inj. 1, 2-5 years | 7.04 [5.67 to 8.74] | 7.74 [5.60 to 10.7]
  Serotype 4; 28 days Post-Inj. 1, 2-5 years: number analyzed (Participants) | 95 | 48
  Serotype 4; 28 days Post-Inj. 1, 2-5 years | 114 [74.0 to 176] | 8.43 [5.97 to 11.9]
  Serotype 4; Pre-Inj. 2, 2-5 years: number analyzed (Participants) | 93 | 46
  Serotype 4; Pre-Inj. 2, 2-5 years | 22.3 [16.0 to 31.0] | 7.64 [5.53 to 10.6]
  Serotype 4; 28 days Post-Inj. 2, 2-5 years: number analyzed (Participants) | 92 | 45
  Serotype 4; 28 days Post-Inj. 2, 2-5 years | 200 [166 to 240] | 8.22 [5.76 to 11.7]
  Serotype 4; Pre-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 44
  Serotype 4; Pre-Inj. 3, 2-5 years | 39.4 [29.5 to 52.8] | 7.97 [5.69 to 11.2]
  Serotype 4; 28 days Post-Inj. 3, 2-5 years: number analyzed (Participants) | 90 | 43
  Serotype 4; 28 days Post-Inj. 3, 2-5 years | 176 [143 to 217] | 9.37 [6.35 to 13.8]
  Serotype 1; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 99 | 49
  Serotype 1; Pre-Inj. 1, 6-11 years | 17.4 [11.4 to 26.6] | 31.0 [16.1 to 59.6]
  Serotype 1; 28 days Post-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 47
  Serotype 1; 28 days Post-Inj. 1, 6-11 years | 41.5 [25.5 to 67.5] | 26.7 [14.2 to 50.0]
  Serotype 1; Pre-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 1; Pre-Inj. 2, 6-11 years | 27.4 [17.2 to 43.6] | 33.9 [17.2 to 66.9]
  Serotype 1; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 1; 28 days Post-Inj. 2, 6-11 years | 165 [122 to 222] | 32.4 [16.6 to 63.2]
  Serotype 1; Pre-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 1; Pre-Inj. 3, 6-11 years | 63.2 [40.5 to 98.7] | 37.2 [18.4 to 75.4]
  Serotype 1;28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 1;28 days Post-Inj. 3, 6-11 years | 207 [152 to 283] | 34.7 [17.4 to 69.1]
  Serotype 2; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 99 | 49
  Serotype 2; Pre-Inj. 1, 6-11 years | 8.57 [6.67 to 11.0] | 9.32 [6.48 to 13.4]
  Serotype 2; 28 days Post-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 47
  Serotype 2; 28 days Post-Inj. 1, 6-11 years | 18.8 [13.5 to 26.2] | 8.40 [6.07 to 11.6]
  Serotype 2; Pre-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 2; Pre-Inj. 2, 6-11 years | 13.3 [9.80 to 18.0] | 8.50 [6.14 to 11.8]
  Serotype 2; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 2; 28 days Post-Inj. 2, 6-11 years | 26.5 [19.7 to 35.7] | 7.92 [5.82 to 10.8]
  Serotype 2; Pre-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 2; Pre-Inj. 3, 6-11 years | 14.1 [10.5 to 19.0] | 7.85 [5.75 to 10.7]
  Serotype 2; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 2; 28 days Post-Inj. 3, 6-11 years | 25.0 [19.4 to 32.3] | 7.55 [5.59 to 10.2]
  Serotype 3; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 99 | 49
  Serotype 3; Pre-Inj. 1, 6-11 years | 14.4 [10.3 to 20.2] | 21.8 [12.8 to 37.1]
  Serotype 3; 28 days Post-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 47
  Serotype 3; 28 days Post-Inj. 1, 6-11 years | 45.6 [31.0 to 67.1] | 18.3 [11.0 to 30.4]
  Serotype 3; Pre-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 3; Pre-Inj. 2, 6-11 years | 25.6 [17.8 to 37.0] | 19.2 [11.9 to 31.1]
  Serotype 3; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 3; 28 days Post-Inj. 2, 6-11 years | 126 [98.6 to 162] | 19.1 [11.8 to 30.8]
  Serotype 3; Pre-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 3; Pre-Inj. 3, 6-11 years | 35.6 [25.3 to 50] | 15.8 [10.2 to 24.6]
  Serotype 3; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 3; 28 days Post-Inj. 3, 6-11 years | 91.3 [73.0 to 114] | 16.7 [10.7 to 26.0]
  Serotype 4; Pre-Inj. 1, 6-11 years: number analyzed (Participants) | 99 | 49
  Serotype 4; Pre-Inj. 1, 6-11 years | 8.03 [6.23 to 10.3] | 8.43 [5.94 to 12.0]
  Serotype 4; 28 days Post-Inj. 1, 6-11 years: number analyzed (Participants) | 98 | 47
  Serotype 4; 28 days Post-Inj. 1, 6-11 years | 68.2 [45.6 to 102] | 7.28 [5.36 to 9.88]
  Serotype 4; Pre-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 4; Pre-Inj. 2, 6-11 years | 20.3 [14.6 to 28.1] | 7.82 [5.90 to 10.3]
  Serotype 4; 28 days Post-Inj. 2, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 4; 28 days Post-Inj. 2, 6-11 years | 126 [96.3 to 164] | 7.44 [5.63 to 9.83]
  Serotype 4; Pre-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 47
  Serotype 4; Pre-Inj. 3, 6-11 years | 39.0 [28.6 to 53.2] | 7.06 [5.37 to 9.29]
  Serotype 4; 28 days Post-Inj. 3, 6-11 years: number analyzed (Participants) | 96 | 46
  Serotype 4; 28 days Post-Inj. 3, 6-11 years | 125 [98.9 to 157] | 7.82 [5.79 to 10.6]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from Day 0 (post-vaccination) up to 28 days post-injection 3. Solicited Reaction (SR) data were collected within 7 and 14 days after vaccination. Serious adverse event (SAE) data were collected throughout the study.
Description: Analysis was performed on Safety Analysis Set. A solicited reaction is an AE that is prelisted in the electronic case report form (eCRF) and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and time to onset) prelisted in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | CYD Dengue Vaccine Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/99
Serious Adverse Events (participants affected / at risk) | 2/199 | 4/99
Other Adverse Events (participants affected / at risk) | 71/199 | 29/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=199) | Control Group (N=99)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vascular purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epiphyseal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=199) | Control Group (N=99)
Injection site Pain; Post-injection 1, All participants (General disorders) | 41 (41) | 17 (17)
Injection site Erythema; Post-injection 1, All participants (General disorders) | 15 (15) | 4 (4)
Injection site Swelling; Post-injection 1, all participants (General disorders) | 11 (11) | 5 (5)
Injection site Pain; Post-injection 2, All participants (General disorders) | 37/188 (37) | 16/92 (16)
Injection site Pain; Post-injection 3, All participants (General disorders) | 33/186 (33) | 29/90 (29)
Injection site Erythema; Post-injection 3, All participants (General disorders) | 8/186 (8) | 10/90 (10)
Injection site Swelling; Post-injection 3, All participants (General disorders) | 6/186 (6) | 8/90 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.